CLINICAL TRIAL: NCT05373160
Title: Determination of Age- and Gender-specific Reference Values of Different Functional Tests With or Without Cognitive Dual-task in Young Adults
Brief Title: Reference Values of Different Functional Tests With or Without Cognitive Dual-task in Young Adults
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cigdem Emirza, Research Assistant, Istanbul Bilgi University
Other Study IDs: qH25cGJv
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Dual-task; Functional Test
Keywords: dual-task; functional test; healthy young; reference value
MeSH Terms: interventions — Outcome Assessment, Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy young group: Individuals who are 18-35 years, did not diagnosed with musculoskeletal disorder, and volunteers
  Interventions: Other: Assessment study

INTERVENTIONS:
Other: Assessment study — Assessment of functional tests with and without dual tasks

SUMMARY:
In this study, reference values for the five basic functional tests that are commonly used, with and without the addition of dual-task activity, will be determined. It will be ensured that healthy normative data that researchers and clinicians can compare in determining the effects in different pathologies by using easy-to-perform evaluations. The aim of this study is to determine the reference values performed with and without dual-task of the five functional tests for young adults according to age and gender by considering the interaction between both mobility and cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years
* Individuals who were not diagnosed with musculoskeletal disorder
* Volunteers

Exclusion Criteria:

* Using an assistive device for walking
* Having cognitive problems
* Individuals who had undergone lower extremity surgery due to musculoskeletal problems in the last six months
* Body mass index greater than 30 kg/m2

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young people
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test without dual task | Baseline
  The test measures the time (in seconds) will taken by a participant to stand up from a chair, walk a distance of 3 m, turn, walk back to the chair, and sit down. To perform the test, the participants will sit on a chair, placing his/her back against the backrest and resting his/her arms on armrests. On the instruction "Go", the participants will rise up from a chair, walk to a line/block on the floor 3 m away, turn around, return, and sit back on a chair.
4 Meter Gait Speed Test without dual task | Baseline
  The participant will walk briskly through the 1-meter "test" zone for acceleration, the central 4-meter "test" zone, and the 1-meter deceleration zone. Time starts with the first leg after the 0 meter line and time is stopped with the first leg after the 4 meter line. In this test, the result is recorded in meters per second (m/s).
10 Meter Walk Test without dual task | Baseline
  In this test, the participant will walk at the best possible speed in a pre-measured 10-meter area. The time starts when the participant's foot is on the starting line and ends when they cross the finish line. In this test, the result is recorded in total seconds.
Timed 25-Foot Walk Test without dual task | Baseline
  The participant walks the distance of 7.62 meters as fast as possible but without running. The time to complete the distance will recorded in seconds.
1 min-Sit-to-Stand Test without dual task | Baseline
  Participants put their hands on their hips and they had to stand up and sit down completely and as many times as possible from a chair (height = 46 cm) without arm rests during one minute. Participants are not allowed to use their arms as support. The number of sit-ups performed during 1 minute will recorded.
Timed Up and Go Test with dual task | Baseline
  The test measures the time (in seconds) will taken by a participant to stand up from a chair, walk a distance of 3 m, turn, walk back to the chair, and sit down. To perform the test, the participants will sit on a chair, placing his/her back against the backrest and resting his/her arms on armrests. On the instruction "Go", the participants will rise up from a chair, walk to a line/block on the floor 3 m away, turn around, return, and sit back on a chair. The participants will perform with dual task. This dual task will be to say the names of animals.
4 Meter Gait Speed Test with dual task | Baseline
  The participant will walk briskly through the 1-meter "test" zone for acceleration, the central 4-meter "test" zone, and the 1-meter deceleration zone. Time starts with the first leg after the 0 meter line and time is stopped with the first leg after the 4 meter line. In this test, the result is recorded in meters per second (m/s). The participants will perform with dual task. This dual task will be counting down the months of the year starting from December.
10 Meter Walk Test with dual task | Baseline
  In this test, the participant will walk at the best possible speed in a pre-measured 10-meter area. The time starts when the participant's foot is on the starting line and ends when they cross the finish line. In this test, the result is recorded in total seconds. The participants will perform with dual task. This dual task will be counting numbers back from 100 by threes.
Timed 25-Foot Walk Test with dual task | Baseline
  The participant walks the distance of 7.62 meters as fast as possible but without running. The time to complete the distance will recorded in seconds. The participants will perform with dual task. This dual task will be counting numbers back from 100 by sevens.
1 min-Sit-to-Stand Test with dual task | Baseline
  Participants put their hands on their hips and they had to stand up and sit down completely and as many times as possible from a chair (height = 46 cm) without arm rests during one minute. Participants are not allowed to use their arms as support. The number of sit-ups performed during 1 minute will recorded. The participants will perform with dual task. This dual task will be counting city names.

CONTACTS AND LOCATIONS:
Overall Officials: Yildiz Analay Akbaba, PT, phD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahman HB, Berglund L, Cedervall Y, Giedraitis V, McKee KJ, Rosendahl E, Aberg AC. Timed "Up & Go" Dual-Task Tests: Age- and Sex-Specific Reference Values and Test-Retest Reliability in Cognitively Healthy Controls. Phys Ther. 2021 Oct 1;101(10):pzab179. doi: 10.1093/ptj/pzab179. PMID 34272869